CLINICAL TRIAL: NCT03634046
Title: Efficacy and Safety of Percutaneous Transforaminal Endoscopic Discectomy Versus Radiofrequency Ablation in the Treatment of Lumbar Intervertebral Disc Herniation: a Case-control Study
Brief Title: PTED Versus Radiofrequency Ablation for Lumbar Disc Herniation
Acronym: PTED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2016T-15; 81371987 (Other Grant/Funding Number: Natural Science Foundation of China)
Record Dates: First submitted 2018-07-17; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Lumbar Disc Herniation; Chronic Low Back Pain
Keywords: Lumbar Disc Herniation; Low Back Pain; Percutaneous Transforaminal Endoscopic Discectomy; Radiofrequency Ablation
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Subjects were recruited comparatively into two groups (percutaneous transforaminal endoscopic discectomy (PTED) group and Radiofrequency Ablation (RA) group). The follow-up time points are 7 days, 1 month, 6 months and 12 months post-operation in both groups, respectively.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor do not know all the information about the data origin and the group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTED group (Experimental): Percutaneous transforaminal endoscopic discectomy (PTED). Use German Joimax company production of intervertebral foramen mirror operation system, the prone position, by preoperative X-ray locating the skin into the needle point, intervertebral level away from the spine line 8 ~ 10 cm, 18 g needle insertion, the Kambin security triangle directly through the middle of pathological changes of intervertebral disc. After the success of the puncture, remove the needle core, injection of contrast agent, methylene blue (9:1) mixture disk imaging, replace the godet, slight rotation step by step to insert the expansion sleeve, X-ray perspective to determine work under the correct position. Radiofrequency ablation is used to form nucleus pulposus and fibrous ring and stop bleeding.
  Interventions: Procedure: Percutaneous transforaminal endoscopic discectomy; Procedure: Radiofrequency ablation
- RA group (Active Comparator): Radiofrequency ablation (RA). Patients in prone position, local infiltration anesthesia, the puncture point for lesion clearance level, is apart from the spine line distance is 8 to 10 cm, in the perspective of the C-shaped arm X-ray machine; After the puncture needle was reached, the needle core was removed and the radiofrequency head was pierced through the puncture channel to the nucleus pulposus. In accordance with the method of melt into the shrinking exit, the intensity of the treatment by band 2, increased to 3 file again, according to the needle round mouth of 2, 4, 6, 8, 10, 12 o'clock to this process is repeated six times.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Percutaneous transforaminal endoscopic discectomy — The same as the descriptions in experimental group.
  Arms: PTED group
Procedure: Radiofrequency ablation — The same as the descriptions in active comparator group.

SUMMARY:
Lumbar disc herniation (LDH) is a common and frequently-occurring disease giving rise to low back pain and (or) leg pain. There are about 1.5 million people with LDH-related pain, accounting for 10% of outpatients each year in China. The mechanism of LDH-related pain is that the degeneration causes the protrusion of the intervertebral disc directly to the lower lumbar nerve root or spinal cord, and the chemical stimulation plays a key role in it. Currently, LDH treatments are mainly divided into conservative treatment, surgical treatment and minimally invasive treatment. The minimally invasive technique is a new technology that has been arising in recent years, with small wound, little bleeding and quick recovery. It mainly includes collagenase dissolving, laser decompression, radiofrequency ablation, etc. Intervertebral disc radiofrequency ablation is an early application of minimally invasive technique with a wide range of applications in a long time. The percutaneous transforaminal endoscopic discectomy (PTED) is a new technique, which is applied in clinics with shorter time, and the implementation and efficacy of the technique need to be further discussed. A case-control clinical trial is designed to compare the efficacy and safety of PTED with radiofrequency ablation in the treatment of LDH. Main outcome is Visual Analogue Scale for leg pain, secondary outcomes are Oswestry disability index, quality of life assessment, Burns Depression Checklist, recovery rate, complications, operation time and radiation exposure time, etc. The follow-up time points are 7 days, 1 month, 6 months and 12 months post-operation.

DETAILED DESCRIPTION:
Please see the Eligibility Criteria or Outcome Measures sections.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar intervertebral disc herniation has been treated with conservative treatment of > for 3 months, or can only temporarily improve symptoms to relieve pain, but can not be maintained for a long time, aged between 18 and 60;
* The symptoms and signs of lumbar intervertebral disc herniation are obviously consistent with those of CT or MRI;
* The protrusion size was < 8.0mm, and imaging examination showed the protrusion of intervertebral disc, mild or moderate protrusion, without calcification, dissociation, and osseous spinal stenosis;
* Patients have a strong desire to treat, and understand radiofrequency thermal coagulation ablation and intervertebral endoscopic treatment of possible risk patients;
* Conservative treatment is ineffective and the surgical treatment is rejected.

Exclusion Criteria:

* The non-inclusion or prominent calcification, dissociation, dissociation and consolidation of vertebral canal stenosis or caudal syndrome in the rupture of the fibrous ring and posterior longitudinal ligament;
* Patients with spinal fractures, tumors and intervertebral discs have skin infections that affect the puncture;
* The combination of mental illness or cognitive dysfunction;
* Patients with serious diseases such as active tuberculosis or heart, lung, liver and kidney;
* Abnormal bleeding or coagulation function caused by various reasons;
* Menstrual period and lactation period;
* No informed consent is signed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-26 (Estimated)

PRIMARY OUTCOMES:
Changes on the Visual Analogue Scale for Leg Pain | Baseline, 7 days, 1 month, 6 months and 12 months post-operation.
  Draw a line of 100 mm on the paper, the end of the horizontal line is 0, indicating no pain; The other end is 10, which is a very serious pain; The middle section shows varying degrees of pain. Let the patient draw a mark on the horizontal line to indicate the extent of the pain.

SECONDARY OUTCOMES:
Changes on the Oswestry Disability Index (ODI) | Baseline, 7 days, 1 month, 6 months and 12 months post-operation.
  The ODI was developed by Fairbank to assess functional impairment. There are 10 questions evaluating various daily activities of this scale and 6 options for each question between 0-5. In this scale, the degree of clinical pain severity, personal care, lifting, walking, sitting, standing, sleeping, social life, travel and change degree of the pain are questioned. The minimum score taken from the scale is 0, the maximum score is 50. 0-4 points mean there is no disability, 5-14 points are mild, 15-24 points are moderate, 25-30 points are severe and 35-50 points are considered to be complete functional disability.
Changes on 36-Item Short-Form Quality of Life Questionnaire (SF-36) | Baseline, 7 days, 1 month, 6 months and 12 months post-operation.
  Short Form-36 (SF-36) will assess the health-related quality of life of individuals. The form consists of a total of 36 articles which can be filed by the patient. The scale consists of 8 subscales related to health. Physical function (10 articles), social function (2 articles), role limitations due to physical problems (3 articles), role limitations due to emotional problems (3 articles), mental health (5 articles), fitness (4 articles), pain (2 articles), general health [general overview point (5 articles) and health change (1 article)]. The scores from each subscale range from 0-100. 0 indicates the worst condition and 100 the best health condition. The SF-36 is suitable for personal evaluation, and can be applied to people over 14 years of age or face to face computerized or trained personnel.
Changes on Burns Depression Checklist | Baseline, 7 days, 1 month, 6 months and 12 months post-operation.
  List of evaluation index for Burns Depression (Burns' Checklist, business data catalog) and business data catalog including 15 items, each item has four degree options (no, mild, moderate, severe) and, in turn, score of 0, 1, 2, 3 points, and then calculate a score (i.e., Depression index), symptom is heavier, the higher the score. Depression rating: 11 ~ 20 points, mild; 21 ~ 30 minutes, moderate; 31 ~ 45 minutes, heavy. For moderate or severe depression, you need to be treated by a psychiatrist and not be involved in this trial.
Changes on the Visual Analogue Scale for Back Pain | Baseline, 7 days, 1 month, 6 months and 12 months post-operation.
  The pain intensity in the back will be measured on a scale from 0 (no pain) to 100 mm (worst imaginable pain).
Complications | through study completion, up to 1year of follow-up.
  A systematic assessment of complications (including wound infection, deep venous thrombosis, urine tract infection, hematoma, and progressive neurological deficit) will be recorded out by the surgeon and research nurse, and these data are to be extracted from the patient chart. Moreover, surgeons will be asked for perioperative complications.
Perceived recovery | Baseline, 7 days, 1 month, 6 months and 12 months post-operation.
  To measure the perceived recovery a seven-point Likert scale will be used. The score on this scale vary from 'completely recovered' to 'worse than ever'.

CONTACTS AND LOCATIONS:
Overall Officials: Yingang Zhang, MD, Principal Investigator — First Affiliated Hospital, Medical College of Xi'an Jiaotong University
Locations (1):
- FirstXianJiaotongU, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No